CLINICAL TRIAL: NCT06913998
Title: The Prevalence and Impacts of Nudix Hydrolase 15 (NUDT15) Gene Variants in Taiwanese Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202309124RINB
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases; Neutropenia; Nudt15 Deficiency
MeSH Terms: conditions — Inflammatory Bowel Diseases; Neutropenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will include participants who were diagnosed with inflammatory disease and followed up at National Taiwan University Children's Hospital. The investigators will check the NUDT15 gene test, if the participant agrees to do an additional blood test. The result of the gene test will be analyzed and compared with other clinical data.

DETAILED DESCRIPTION:
In inflammatory bowel disease (IBD), thiopurines play an important role in maintenance of steroid-free remission but possess risk of life-threatening neutropenia, which is associated with gene variants of NUDT15 in Asians. In order to better incorporate thiopurines in clinical practice, the investigators aim to summarize the prevalence and impacts of NUDT15 variation in IBD in Taiwan. The study will include participants who were diagnosed with inflammatory disease and followed up at National Taiwan University Children's Hospital. The investigators will check the NUDT15 gene test, if the participant agrees to do an additional blood test. The result of the gene test will be analyzed and compared with other clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with inflammatory bowel disease.

Exclusion Criteria:

* Participants who refused to have blood test for NUDT15 gene evaluation.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study included participants who are diagnosed with inflammatory bowel disease at National Taiwan University Children's Hospital and agree to have blood test for NUDT15 gene evaluation.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Neutropenia | 2 years
  Neutropenia is defined as absolute neutrophil count <1500/microL, and severe neutropenia is defined as absolute neutrophil count <500/microL.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan